CLINICAL TRIAL: NCT06759311
Title: Clinical Assessment of Two Different Minimal Invasive Techniques in Caries Removal of Primary Teeth (Randomized Control Clinical Trial)
Brief Title: Two Different Minimal Invasive Techniques in Caries Removal of Primary Teeth
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant Lecturer of Dental Public Health and biostatistical consultanat, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 235-25-08-2024
Record Dates: First submitted 2024-12-23; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Dental Caries in Children
Keywords: Minimal Invasive Dentistry

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ART (Active Comparator)
  Interventions: Other: ART
- Brix 3000 (Experimental)
  Interventions: Other: Brix 3000
- Carie Move (Experimental)
  Interventions: Other: Carie Move
- Smart Bur (Experimental)
  Interventions: Other: Smart Bur

INTERVENTIONS:
Other: ART — The restorative procedure performed in relative isolation and without the use of anesthesia consisted of removal of the carious tissue using hand instrument excavators and dentin
  Arms: ART
Other: Brix 3000 — Brix 3000 gel will be applied to the caries lesion using a spoon excavator** leaving gel according to the manufacturer's instructions. After 2 minutes, the gel will turn from translucent green colour to cloudy after the gel removal.
  Arms: Brix 3000
Other: Carie Move — Carie-Move gel will be applied to the caries lesion according to the manufacturer's instructions at second visit in the same child. After 30 second the gel will be removed.
  Arms: Carie Move
Other: Smart Bur — Removal of carious dentin will be carried out employing smart bur II mounted on a low-speed handpiece without water spray. Caries removal will be proceeded until the smart bur II becomes dull after repeated contact with healthy dentin (21) (figure 3)
  Arms: Smart Bur

SUMMARY:
Pain control during dental treatments is the most challenging situations that face the pediatric dentist especially in young and fearful or anxious child. Minimal invasive approach for caries removal includes many techniques to remove caries either by dental excavators, rotatory burs, atraumatic restorative treatment (ART), chemo-mechanical caries removal and smart bur.

ELIGIBILITY:
Inclusion Criteria:

* Each child has three teeth with carious cavity enough for insertion of hand instruments
* Positive or definitely positive child behaviour according to the Frankl Behaviour Scale (FBS)
* Caries lesion in dentin of primary teeth

Exclusion Criteria:

* Negative" or "definitely negative" child behaviour according to the FBS.
* Presence of sign and symptoms of pulp lesion

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-02-20 (Estimated)

PRIMARY OUTCOMES:
pain scores | Immediately after the intervention
  Wong-Baker Faces Pain Rating Scale (WBFPS) Presents 6 faces with increasing degrees of pain from left to right. Each face was attributed a scale from 0 to 10 indicated onthe scale.
  Children were asked to choose the face that best describe his or her pain.
caries removal time | During procedure
  The total working time required for caries removal will be recorded in minutes using a stopwatch
Caries removal efficacy | Immediately after the intervention
  The caries removal criteria:
  0 Caries removed completely
  1. Caries noticed at the base of the cavity
  2. Caries noticed at the base and/or one wall of the cavity
  3. Caries noticed at the base and/or two walls of the cavity
  4. Caries noticed at the base and/or more than two walls of the cavity
  5. Caries noticed at the base, walls and margins of the cavity.

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinic of Pediatric dentistry, Faculty of dentistry, pharos University, Egypt, Alexandria, Egypt